CLINICAL TRIAL: NCT05217134
Title: Sacral Anesthetic Block During Labor Analgesia With a With a 27-G Whitacre Spinal Needle - Dural Puncture Epidural Technique vs Standard Epidural Technique: a Randomized Controlled Study.
Brief Title: Sacral Spread of Sensory Block After Dural Puncture Epidural Technique Compared With Epidural for Labour Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4294
Record Dates: First submitted 2021-11-29; First posted 2022-02-01 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Labor Pain; Analgesia
Keywords: Dural Puncture Epidural Analgesia; Sacral pain
MeSH Terms: conditions — Labor Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dural Puncture Epidural Analgesia (DPEA) (Experimental): A 27-Whitacre spinal needle puncture will be performed with confirmation of LCR return, before the introduction of epidural catheter.
  Interventions: Procedure: DPEA
- Epidural Analgesia (EA) (No Intervention): Standard epidural anesthesia wil be performed.

INTERVENTIONS:
Procedure: DPEA — Dural puncture with 27 G Whitacre needle
  Arms: Dural Puncture Epidural Analgesia (DPEA)

SUMMARY:
Neuraxial labor analgesia is a very widely used technique for labor pain relief with a high efficacy and safety. EA (Epidural analgesia) can guarantee a proper control of pain in 95-100% of cases in the first stage of labor, but in the second stage his efficacy is not always adequate. DPEA (Dural Puncture Epidural Analgesia) is a variation of the conventional EA and technically a modified version of the CSE (Combined Spinal Epidural) analgesia.

When compared with the traditional EA, DPEA showed satisfying, effective and fast control of labor pain, no motor block and less need for anesthetic boluses given through the epidural catheter when the maintenance of analgesia was guaranteed with manual top-ups, as well as less request for extra boluses of anesthetic when PIEB (Programmed Intermittent Epidural Boluses) was chosen for the maintenance of analgesia. Studies proved that DPEA is a safe technique and no statistically significant incidence of side effects for mothers and fetuses was observed.

The hypothesis of this study is that a DPEA performed with a 27 G Whitacre spinal needle can especially improve the spread in the sacral region.

The primary outcome of this study is to evaluate whether the DPEA performed with a 27-G Whitacre spinal needle is more effective in ensuring satisfying analgesia as a result of a better sacral analgesic spread, compared to the traditional EA.

DETAILED DESCRIPTION:
Labor pain is acute pain, with a sudden onset, limited duration, high intensity and an evolving character consisting of a visceral and a somatic component1. Many dermatomes are involved, unlike other pain syndromes.

In the first stage of labor, pain is caused by the contraction of the uterine fibers and by the stretching and dilation of the cervix and the lower uterine segment. When labor proceeds towards the active phase of the first stage, corresponding to a dilation of 3-4 cm, the pain becomes more severe, and extends to the contiguous dermatomes T10 and L1. The pain generated at this moment is visceral, dull, indistinct, difficult to locate, "referred" to skin areas far from the site of pain stimulation and most of the time as "back pain". When the uterine cervix is fully dilated, the second stage of labor begins: the pain is due to the distension and stretching of the perineal structures in conjunction with fetal progression. This late pain originates from the perineum (deep somatic pain) and is conducted by type A-delta and C somatic myelin fibers, that through the pudendal nerves reach the posterior horns of the spinal cord via the posterior roots of the 2nd, 3rd and 4th sacral nerve.

Currently, neuraxial analgesia is a very widely used technique for labor pain relief with a high efficacy and safety. Neuraxial analgesia is administered through:

* continuous or intermittent epidural block
* continuous or single shot spinal or subarachnoid block
* combined spinal-epidural block (CSE). DPEA (Dural Puncture Epidural Analgesia) is a modified version of the CSE analgesia technique and at the same time a combination of CSE and EA (Epidural Analgesia). Despite the similarities, the management of labor analgesia with these techniques is profoundly different. DPEA does not allow the same rapid onset of CSE analgesia, since the administration of the intrathecal dose is omitted, but the induction and maintenance of analgesia are guaranteed by the epidural catheter as in the standard AE.

EA (Epidural analgesia) can guarantee a proper control of pain in 95-100% of cases in the first stage of labor, but in the second stage his efficacy is not always adequate.

DPEA is a variation of the conventional EA and technically a modified version of the CSE analgesia.

It is performed by making an intentional puncture of the dura mater with a spinal needle, that is inserted in the Tuohy needle previously placed in the epidural space, without any administration of intrathecal medications.

If compared with the traditional EA, DPEA showed satisfying, effective and fast control of labor pain, no motor block and less need for anesthetic boluses given through the epidural catheter when the maintenance of analgesia was guaranteed with manual top-ups, as well as less request for extra boluses of anesthetic when PIEB (Programmed Intermittent Epidural Boluses) was chosen for the maintenance of analgesia.

Studies proved that DPEA is a safe technique and no statistically significant incidence of side effects for mothers and fetuses was observed.

DPEA can't provide the same analgesia's fast onset of the CSE, as no medications are given in the intrathecal space7-8, but authors agree that DPEA produces a better quality of labor analgesia compared with the EA.

The advantages of the DPEA include: less cases of wrong placement of the epidural catheter because of the confirmation given by the cerebrospinal fluid return, more hemodynamic stability, less risk of unilateral block and consequent manipulation and replacement of the epidural catheter, but most of all, the spontaneous translocation of a certain amount of anesthetic from the epidural to the intrathecal space through the little hole made intentionally in the dura mater could improve the strength of the analgesia both in the first and in the second stage of labor.

After the the acquisition of informed consent, all the nulliparous, singleton, vertex presenting pregnant women in labor between the 36th and 42nd gestational week and with less than 5 cm cervical dilation will be randomized according to a computer-generated random number sequence to receive DPEA or EA.

For all pregnant women, an 18 G intravenous access will be positioned before performing the neuro-axial technique and fluid therapy with Ringer Lactate 1000 ml will be started. Non-invasive multiparametric monitoring will include pulse oximetry, NIBP (Non Invasive Blood Pressure) and CTG (Cardiotocography).

The epidural space will be identified in both groups with a Tuohy 18 G needle using the loss of resistance technique to saline with liquid syringe and the spinal needle (Whitacre 27 G) inserted using the "needle through needle" technique. In patients randomized to receive a DPEA, a single spinal needle puncture will be performed with confirmation of LCR return, while in the EA group no hole will be drilled in the dura mater.

A 20 G multi-orifice epidural catheter will be inserted 5 cm inside the peridural space. After negative suction test for blood and LCR, an initial dose of 15 ml of ropivacaine 0.1% + sufentanil 0,5 mcg /ml will be administered through the peridural catheter. The maintenance of analgesia will be guaranteed through a PIEB machine, that will give to the patient every hour a single bolus of 10 ml of ropivacaine 0,1% + sufentanil 0,5 mcg/ml. In case of insufficient analgesia (breakthrough pain, VAS > 4) a rescue dose of 10 ml of 0.13% ropivacaine will be administered.

A rescue dose of 10 ml of 0.15% ropivacaine will be used to treat breakthrough pain at complete cervical dilatation.

The sample will be described in its clinical and demographic characteristics through descriptive statistics techniques. In particular, the qualitative variables will be represented with absolute and percentage frequency tables; continuous quantitative variables with normal distribution, with mean, standard deviation or 95%confidence interval; non-normal variables will be represented with minimum, maximum and mean.

Missing data will be presented in the form of n (%). The normality of continuous variables will be verified with the Shapiro-Wilk test and will be adopted opportune modifications when requested. The variance's similarity will be verified with the sd test. The primary objective will be assessed by comparing the incidence of the sensitive perineal block in two groups of patients at fixed time points, reporting risk ratios, 95% confidence interval and p values through the Chi square test or the Fisher test for estimated < 5 frequencies. The same method will be used to evaluate the secondary outcomes' incidence. To compare the differences between continuous quantitative variables with a normal distribution the Student t-test for independent samples will be applied. For variables with non-normal distribution the Mann-Whitney non parametric test for independent samples will be performed. A p value <0.05 will be considered significant.

All analyzes will be performed with the statistical software STATA IC 15.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous;
* 36 - 42 gestational week;
* active stage of labor;
* less than 5 cm cervical dilatation.

Exclusion Criteria:

* < 18 years;
* ASA > 2;
* refusal of informed consent;
* known fetal pathologies;
* conditions that contraindicate the execution of neuro axial analgesia techniques;
* uterine anomalies or previous uterine surgery;
* severe obesity;
* twin pregnancy;
* non-vertex fetal presentation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients
Enrollment: 108 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of sensitive block through a pin-prik test in lumbar and sacral dermatomes. | 20 minutes after completion of anesthesia.
  Efficacy of sacral anesthetic block through a pin-prik test (0= no sensitive block, 2= complete block) in lumbar and sacral dermatomes: stimulation of the inguinal ligament (L1), the anterior portion of the thigh (L2), the medial surface of the knee (L3), the medial malleolus (L4), the back of the foot in the space between the first two metatarsal rays (L5), the lateral surface of the heel (S1) and the medial popliteal fossa (S2).

SECONDARY OUTCOMES:
Change of pain relief | 10 minutes, 20 minutes, 30 minutes and then every 1 hour after completion of anesthesia.
  Visual Analogue Pain Score (0=no pain, 10=the worst imaginable pain) throughout the labor
Supplemental analgesia requirement | 20 minutes after delivery.
  Total volume of anesthetic given as a rescue dose to treat episodes of breakthrough pain.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Policlinico Agostino Gemelli, Rome
  - Luciano Frassanito, Rome

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gunaydin B, Erel S. How neuraxial labor analgesia differs by approach: dural puncture epidural as a novel option. J Anesth. 2019 Feb;33(1):125-130. doi: 10.1007/s00540-018-2564-y. Epub 2018 Oct 6. PMID 30293143
- [Result] Shmueli A, Salman L, Orbach-Zinger S, Aviram A, Hiersch L, Chen R, Gabbay-Benziv R. The impact of epidural analgesia on the duration of the second stage of labor. Birth. 2018 Dec;45(4):377-384. doi: 10.1111/birt.12355. Epub 2018 May 22. PMID 29790194
- [Result] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707
- [Result] Contreras F, Morales J, Bravo D, Layera S, Jara A, Riano C, Pizarro R, De La Fuente N, Aliste J, Finlayson RJ, Tran DQ. Dural puncture epidural analgesia for labor: a randomized comparison between 25-gauge and 27-gauge pencil point spinal needles. Reg Anesth Pain Med. 2019 May 22:rapm-2019-100608. doi: 10.1136/rapm-2019-100608. Online ahead of print. PMID 31118278
- [Result] Cappiello E, O'Rourke N, Segal S, Tsen LC. A randomized trial of dural puncture epidural technique compared with the standard epidural technique for labor analgesia. Anesth Analg. 2008 Nov;107(5):1646-51. doi: 10.1213/ane.0b013e318184ec14. PMID 18931227
- [Result] Thomas JA, Pan PH, Harris LC, Owen MD, D'Angelo R. Dural puncture with a 27-gauge Whitacre needle as part of a combined spinal-epidural technique does not improve labor epidural catheter function. Anesthesiology. 2005 Nov;103(5):1046-51. doi: 10.1097/00000542-200511000-00019. PMID 16249679
- [Result] Song Y, Du W, Zhou S, Zhou Y, Yu Y, Xu Z, Liu Z. Effect of Dural Puncture Epidural Technique Combined With Programmed Intermittent Epidural Bolus on Labor Analgesia Onset and Maintenance: A Randomized Controlled Trial. Anesth Analg. 2021 Apr 1;132(4):971-978. doi: 10.1213/ANE.0000000000004768. PMID 32282386